CLINICAL TRIAL: NCT02639234
Title: A Phase 2 Study of Vigil™ Augmented Autologous Tumor Cell Immunotherapy in Combination With Nivolumab PD-1 Inhibitor for Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Vigil™ + Nivolumab in Advanced Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-122
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Advanced Non-small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer; Lung Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — FANG vaccine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vigil™ + Nivolumab (Experimental): Patients meeting study eligibility criteria will receive doublet therapy comprising of (i) Vigil™ 1 x 10^7 cells by intradermal injection every 2 weeks (for a minimum of 4 and a maximum of 12 doses) and (ii) nivolumab 3 mg/kg by intravenous infusion over 60 minutes every 2 weeks.
  Interventions: Biological: Vigil™; Drug: Nivolumab

INTERVENTIONS:
Biological: Vigil™ — Upon completion of nivolumab infusion, subjects will receive Vigil™, 1.0 x 10^7cells via intradermal injection on Day 1 every 14 days for a minimum of 4 and a maximum of 12 doses depending on quantity of Vigil™ manufactured from surgical specimens.
  Other Names: formerly known as FANG™; bi-shRNAfurin and GMCSF Autologous Tumor Cell Immunotherapy
Drug: Nivolumab — Prior to Vigil™, subjects will receive nivolumab 3 mg/kg by intravenous infusion over 60 minutes on Day 1 every 14 days. If nivolumab is administered beyond 12 months it will be administered off study.
  Other Names: PD-1/PD-L1 checkpoint inhibitor; Opdivo

SUMMARY:
This is an open label phase 2 study to evaluate the combination of Vigil™ and nivolumab in advanced or metastatic NSCLC that is progressive on or after one prior platinum-based systemic therapy. Patients meeting study eligibility criteria will receive Vigil™ every 2 weeks (for a minimum of 4 and a maximum of 12 doses) and nivolumab every 2 weeks. The combination of Vigil™ and nivolumab will demonstrate a higher objective response rate (ORR) than the historical ORR of single agent nivolumab in patients with advanced NSCLC.

DETAILED DESCRIPTION:
This is an open label phase 2 study to evaluate the combination of Vigil™ autologous tumor cell immunotherapy and nivolumab PD-1 inhibitor therapy in patients with advanced or metastatic NSCLC that is progressive on or after one prior platinum-based systemic therapy (ALK or EGFR mutation-targeted therapy should have been received if appropriate mutation present).

Patients undergoing a standard surgical procedure (e.g., tumor biopsy, palliative resection, or thoracentesis of malignant pleural effusion) may elect to have tumor tissue procured for manufacture of Vigil™ vaccine. Patients meeting study eligibility criteria will receive doublet therapy comprising of (i) Vigil™ 1 x 10^7 cells by intradermal injection every 2 weeks for a minimum of 4 and a maximum of 12 doses and (ii) nivolumab 3 mg/kg by intravenous infusion over 60 minutes every 2 weeks. Three to six weeks after tissue procurement has occurred eligibility will be reconfirmed by the study site. Subjects must begin the study regimen within 6 weeks of tissue procurement. Radiological assessment of tumor response will be performed at screening, Cycle 5 (Week 9) and approximately every 2 months thereafter until progressive disease unless the subject is lost to follow-up, withdraws consent for study related procedures, or initiates another cancer therapy. Tumor biopsy for correlative studies should be obtained at tissue procurement and at Cycle 5 (Week 9). Peripheral blood mononuclear cells (PBMC) for correlative studies should be obtained before tumor procurement, and prior to initiation of study therapy on Day 1 at Cycle 1 (Week 1), Cycle 5 (Week 9), Cycle 9 (Week 17) and EOT.

ELIGIBILITY:
Tissue Procurement Inclusion Criteria:

Patients will be eligible for tissue procurement for the Vigil™ manufacturing process, if they meet all of the following criteria:

1. Histologically or cytologically confirmed diagnosis of NSCLC.
2. Age ≥ 18 years.
3. Locally advanced or metastatic disease that is progressive after one prior platinum-based systemic chemotherapy regimen

   1. Adjuvant therapy will count as a line of therapy if administered within 6 months of relapse).
   2. Subjects with EGFR or ALK mutations should also have received appropriate targeted therapy.
4. No systemic therapy, immunologic therapy or investigational therapy within 3 weeks and no radiation therapy within 1 week prior to tumor procurement for vaccine manufacture.
5. Planned standard of care surgical procedure (e.g., tumor biopsy or palliative resection or thoracentesis) and expected availability of a cumulative mass of ~10-30 grams tissue ("golf-ball" size) or pleural fluid estimated volume ≥ 500mL (must be primary tap) for immunotherapy manufacture.
6. At least one area of cancer, not intended for vaccine manufacture, that is measureable by RECIST 1.1 criteria.
7. At least one tumor, not intended for vaccine manufacture, that is considered appropriate for on-treatment biopsy. The same tumor may suffice for both on-treatment biopsy and RECIST 1.1 measurement so long as imaging occurs prior to biopsy.
8. ECOG Performance Status ≤ 1
9. Estimated survival ≥ 6 months.
10. Ability to understand and the willingness to sign a written informed consent document for tissue harvest.

Tissue Procurement Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for tissue procurement for the Vigil™ manufacturing:

1. Any localized anticancer therapy (e.g., radiation, radiofrequency ablation, cryotherapy) to tumor intended for vaccine manufacture unless unequivocal evidence of post-treatment disease progression of the target tumor.
2. Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily for < 30 days duration
3. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
4. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 4 months.
5. Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids.
6. Known history of allergies or sensitivities to gentamicin.
7. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
8. Known HIV or chronic Hepatitis B or C infection.
9. History of pneumonitis or interstitial lung disease.

Study Enrollment Inclusion Criteria:

Patients will be eligible for registration into the trial if they meet all of the following inclusion criteria:

1. Successful manufacturing of at least 4 vials of Vigil™.
2. ECOG Performance Status ≤ 1
3. Estimated survival ≥ 4 months.
4. Disease that is measurable by RECIST 1.1 criteria.
5. Adequate organ function as defined by the following laboratory values:

   Absolute granulocyte count ≥ 1,500/mm3 Absolute lymphocyte count ≥ 500/mm3 Platelets ≥ 75,000/mm3 Hemoglobin ≥ 9 g/dL Creatinine ≤ 1.5x institutional upper limit of normal Total bilirubin ≤ 1.5x institutional upper limit of normal AST(SGOT) and ALT(SGPT) ≤2x institutional upper limit of normal or

   ≤5x institutional upper limit of normal if liver metastases INR / PT and aPTT ≤ 1.5 x ULN (if not using anticoagulants) Immunological Thyroid Stimulating Hormone within institutional limits
6. Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade 2 or better.
7. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
8. Investigator deems the patient to have a tumor appropriate for on-treatment biopsy and patient agrees to provide tissue biopsy at Cycle 5 (Week 9) for correlative studies.
9. Ability to understand and the willingness to sign a written informed protocol specific consent.

Study Enrollment Exclusion Criteria:

In addition to the procurement exclusion criteria, patients will NOT be eligible for study registration and enrollment if meeting any of the following criteria:

1. Any anti-neoplastic therapy between tissue procurement for vaccine manufacture and start of study therapy.
2. Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy.
3. Post-surgery complication that in the opinion of the treating investigator would interfere with the patient's study participation or make it not in the best interest of the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by RECIST 1.1 criteria of Vigil™ plus nivolumab in patients with NSCLC after failure of prior platinum-based chemotherapy | 12 months
  The primary endpoint of ORR is defined as a best response of complete remission (CR) or partial remission (PR) according to RECIST 1.1 as determined by the investigator.

SECONDARY OUTCOMES:
Tolerability and safety profile of Vigil™ combined with nivolumab (all adverse events (CTCAE 4.03), laboratory safety assessments, and physical examination findings) | 12 months
  Safety endpoints include all adverse events (CTCAE 4.03), laboratory safety assessments, and physical examination findings.
Progression-Free Survival (PFS) of study patients treated with Vigil™ and nivolumab | 12 months
  The secondary efficacy endpoint of PFS is the time from randomization to progression according to RECIST version 1.1 or until death from any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Manning, MD, Study Director — Gradalis, Inc.
Locations (3):
- United States (3):
  - Texas Oncology, P.A., Texas Cancer Center, Abilene, Texas
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Cancer Care Northwest, Spokane Valley, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881